CLINICAL TRIAL: NCT04694690
Title: Clinical Performance of Resin Cements in the Adhesion of CAD/CAM Restorations
Brief Title: Clinical Performance of Different Resin Cements
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Simge Canatan, dentist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAD/CAM-hybrid
Record Dates: First submitted 2021-01-02; First posted 2021-01-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Restoration of Posterior Teeth
Keywords: CAD/CAM; Inlay; Onlay; Hybrid ceramic; Adhesive resin cement
MeSH Terms: interventions — RelyX U200; Resin Cements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RelyX U200 Automix Self Adhesive Resin Cement (Experimental): Self Adhesive Resin Cement
  Interventions: Other: Self adhesive resin cement
- G-Cem LinkForce Resin Cement (Active Comparator): Resin Cement system used after surface treatment
  Interventions: Other: Resin cement

INTERVENTIONS:
Other: Self adhesive resin cement — Self adhesive resin cement
  Other Names: RelyX U 200
  Arms: RelyX U200 Automix Self Adhesive Resin Cement
Other: Resin cement — Resin Cement system used after surface treatment
  Other Names: G-Cem LinkForce
  Arms: G-Cem LinkForce Resin Cement

SUMMARY:
The clinical performance of different resin cements in adhesion of hybrid ceramic inlay and onlay restorations produced with CAD/CAM will be evaluated and compared. After obtaining a signed informed consent form from all the patients, all restorations will be placed by a single clinician. All hyrid ceramic restorations (Cerasmart, GC, Tokyo, Japan) will be produced using the same CAD/CAM CEREC Omnicam (Sirona Dental, Bensheim, Germany) system. 70 restorations will be divided into 2 groups: a self adhesive resin cement (RelyX U200 Automix, 3M ESPE, Seefeld, Germany), and an adhesive cement (G-Cem LinkForce, GC, Tokyo, Japan) which is applied after surface treatment (etch&rinse). All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using modified United States Public Health Service (USPHS) criteria after baseline, 6,12, 18, 24, 36 and 48 months. Descriptive statistics will be performed using Friedman test and Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with or without systemic disease
* Patiens older than 18 years old
* Good oral health
* Patients who at least have1 large and deep carious lesion or broken restoration in a vital tooth
* Patients who agreed to participate in the study after being informed about this study

Exclusion Criteria:

* Patient with periodontal disease
* Patients with partial dentures
* Patients with bruxism
* Patients with malooclusion
* Non vital or endodontically treated teeth
* Preparetions under the cemento-enamel junction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | 18 months
  18 months- Modified United States Public Health Service

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided